CLINICAL TRIAL: NCT03913520
Title: Postoperative Outcome of Patients With Congenital Heart Disease Presenting for Non-cardiac Interventions
Brief Title: Outcome of Patients With Congenital Heart Disease
Acronym: OUTCARDIOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/12FEV/072
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Congenital Heart Disease (Other): Undergoing evaluation at 30 days
  Interventions: Other: Outcome research

INTERVENTIONS:
Other: Outcome research — patients will undergo an evaluation of their outcome at 30 days postoperatively

SUMMARY:
Advanced surgical and medical healthcare systems have resulted in an increased prevalence of children and adults with congenital heart disease in Western countries. These patients often necessitate non-cardiac interventions. Previous studies have demonstrated that these patients are at increased risk of morbidity and mortality when presenting for non-cardiac interventions. The aim of this study is to know the prevalence of patients with congenital heart disease presenting for non-cardiac interventions in a tertiary hospital and to determine their outcome.

DETAILED DESCRIPTION:
Previous studies have shown that children and adults presenting with congenital heart disease are at increased risk of morbidity and mortality after non-cardiac interventions. This risk depends on the type of pathology, the age of the patient and the experience of the physicians in charge of these patients.

We sought to determine the prevalence of children and adults with congenital heart disease presenting for non-cardiac interventions and to investigate their outcome.

ELIGIBILITY:
Inclusion Criteria:

* All children and adults with congenital heart disease

Exclusion Criteria:

* Parental or patient refusal
* Patients presenting for cardiac interventions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-28 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of patients with congenital heart disease presenting for non-cardiac interventions in a single-centre tertiary hospital | Intraoperative
  To analyze the exact number of children and adults with congenital heart disease presenting for non-cardiac interventions in a tertiary hospital

SECONDARY OUTCOMES:
To analyze morbidity after non-cardiac interventions in patients with congenital heart disease | 30 days
  Morbidity outcome after non-cardiac interventions
To analyze mortality after non-cardiac interventions in patients with congenital heart disease | 30 days
  Mortality outcome after non-cardiac interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mona MOMENI, MD,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No